CLINICAL TRIAL: NCT06501703
Title: The Impact Of Different Final Irrigation Activation Techniques On Postoperative Pain In Single Rooted Mandibular Premolar Teeth: A Randomized Clinical Trial
Brief Title: The Impact Of Different Final Irrigation Activation Techniques On Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Yasmin Tawfik Mohamed Sobh, Endodontic lecturer, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/832
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Acute Pulpitis With Apical Periodontitis, Postoperative Pain
Keywords: Fanta AF max file, Passive ultrasonic irrigation, Postoperative pain, XP-endo Finisher.
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel double blinded
Who Masked: Participant, Outcomes Assessor
Masking Description: double (participants ,outcome assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- XP Endo finisher (Experimental): technique used for final irrigation in vertical lengthwise movement to the full working length for 1 minute in each canal.
  Interventions: Other: Instruments
- Passive Ultrasonic Irrigation (Experimental): technique used for final irrigation in vertical strokes reaching 2 mm short from the full working length for 1 minute in each canal.
  Interventions: Other: Instruments
- Fanta AF max file (Experimental): technique used for final irrigation in vertical lengthwise movement to the full working length for 1 minute in each canal.
  Interventions: Other: Instruments
- Manual Dynamic agitation (Active Comparator): technique used for final irrigation in Intermittent manual activation for 1 min in up-and-down motion using master gutta percha cone was performed.
  Interventions: Other: Instruments

INTERVENTIONS:
Other: Instruments — instruments used as different techniques in final irrigation after root canal preparation
  Other Names: XP Endo finisher; Passive Ultrasonic Irrigation; Fanta AF max file; Manual dynamic agitation

SUMMARY:
The trial was conducted to assess the impact of passive ultrasonic irrigation, XP endo finisher, AF max file, and manual dynamic agitation on postoperative pain and analgesic consumption at 6 h., 12 h., 24 h., 48 h., 72 h., and a week later on single-rooted lower premolar teeth with acute irreversible pulpitis and apical periodontitis.

DETAILED DESCRIPTION:
Selection of cases:

A total number of sixty-four patients in the 18-40 age range will be enrolled for the study from the outpatient clinic of restorative department of Sinai university (Kantara branch). The selected patients will have a carious pulp exposure that will be selected according to the inclusion and exclusion criteria to participate in this study. the procedure, possible discomfort and benefits will be explained to the patients. Informed consent will be obtained from the patients prior to study which includes root canal treatment in a single visit of single rooted mandibular premolar teeth with carious pulp exposure and symptomatic irreversible pulpitis with apical periodontitis, and both verbal and written consent is advisable. Before initiation of treatment, the whole procedural steps will be explained to the patients. Then the patients will sign an informed consent form.

Sample size:

Sample size calculation was performed using G*Power version 3.1.9.7 based on the results of a previous study) (13). A power analysis was designed to have adequate power to apply a two-sided statistical test to reject the null hypothesis that there is no difference between groups. By adopting an alpha level of (0.05) and a beta of (0.2), i.e. power = 80% and an effect size (d) of (0.55) calculated based on the results of a previous study. The predicted sample size (n) will be (64), i.e., 16 samples per group. To detect for different postoperative pain between groups Patient Selection Criteria Systemically healthy patients with single rooted mandibular premolar teeth with oval canals diagnosed with carious pulp exposure and symptomatic irreversible pulpitis with apical periodontitis will be included in the study. The diagnosis will be based on clinical findings, including pain level and its characteristics, intensity, duration, frequency, and provoking and relieving factors. Intraoral clinical examination had revealed either extensive restoration or a history of significant caries. Digital periapical x-rays had been used to assess the following factors: tooth structure, extensive caries, improper fillings, periapical tissue condition, and periodontal support. Whenever the regular x-rays disclosed participants with doubt of more than one canal, cone beam computed tomography (CBCT) was used to exclude. The inclusion guidelines for individuals' restorable teeth with a normal periodontal score index of less than two were as follows: severe preoperative pain (Vas score 3), discomfort response on biting/mastication or percussion but no mobility. Discomfort response on palpation of surrounding tissue but with no intraoral swelling. The inclusion criteria also include patients who stopped medications for the last 12 hours before the procedure. Additionally, the radiograph showed only normal or slight widening in the periodontal ligament space of the affected root. The exclusion criteria included patients with any serious systemic disease, those under the age of eighteen or incapable of giving informed consent, those over forty, those with severe preoperative pain on biting/mastication or percussion, those with a mandibular premolar involving multiple canals or huge periapical pathosis, open apices, periodontal involvement, retreated cases, sinus tract presence, and swelling of surrounding soft tissues; in addition to those, patients who had been pregnant and allergic patients with local anesthetic agents.(15) All participants will be informed about the study, and their consent will be obtained before treatment. A list for random participant assignment will be generated by a randomization software. This randomization will be performed by an operator not involved in the study. An ethyl chloride cold pulp tester will be used to detect the affected tooth's response and the adjacent and contralateral teeth (used as control) to ensure that the tester will work properly and that the participants responds adequately. The preoperative pain level will be assessed by giving each participant a pain scale chart (VRS) to record the pain level before any intervention. Clinical and radiographic data of each patient will be attached to their clinical notes Preparation of the patient: - Before the preparation and restoration visit, all patients will be subjected to full mouth scaling and will be given proper oral hygiene instruction.

Clinical Steps

The root canal treatment had been completed in one session. The tooth had been anesthetized using a mental nerve block (4% Mepivicaine HCl &1:100,000 adrenaline) and an intraligamentary technique of at least 0.2 ml of the anesthetic solution was injected directly in the periodontal space mesial and distal to the anaesthetized tooth. Following the removal of decay or restorations, an access cavity had been opened. Next, a rubber dam had been applied (Sanctuary Dental Dam Systems, Ipoh, Malaysia). If the patients still complained of pain after giving the anesthesia, around of 0.2 mL of anesthetic solution is injected with adequate pressure to attain intra pulpal anesthesia. Using a 15 K file, canal patency was verified (Dentsply Maillefer). Regarding the electronic apex locator (Root ZX, J. Morita, Tokyo, Japan), the W.L. had been established at the apical constriction and then radiographically verified. Following the manufacturer's recommendations, the root canals had been instrumented through the Protaper Next rotary system (PTN) (Dentsply Maillefer) utilizing an endodontic motor (X Smart, Dentsply Maillefer, Ballaigues, Switzerland) with an adapted torque of 2 Ncm and speed of 300 rpm. The rotary system X4 (40/6%) was worked as the master apical file until it reached the full W.L. Using a 30-gauge side-ventilated needle (NaviTip, Ultradent, UT, USA) that had been placed 2 mm coronal from the W.L. to deliver the irrigating solution. A 2.5% NaOCl solution was injected at a flow rate of 3 ml per minute following each file. The volume of the irrigation delivery during instrumentation was 12 ml. The final active irrigation had been dispensed at a flow rate of 5 mL/minute following endodontic preparation. The time for active irrigation had been standardized in every group to be one minute. The cycles of agitation and replenishment were carried out twice. Based on the final activation irrigation protocol, participants had been separated into four groups as follows:

Group 1: PUI Group 2: XPF Group 3: AF max file Group 4: MDA

For all groups, 5 ml of sterile saline was transported into the canals for one minute to cancel out the carryover effect of NaOCl. After that, 2 ml of 17% ethylene diamine tetraacetic acid (EDTA) solution was passively injected in every group for one minute for smear layer removal. Lastly, 5 ml of sterile saline was delivered for one minute. The canals were dried using aseptic paper points size #40 (Meta Biomed, Cheongju City, Korea). Then, a radiograph was taken using ProTaper® Next Gutta-Percha Points X4# (40/6%) as a master cone. After that, the canals were sealed using the lateral compaction technique. A thick glass ionomer (GI; KetacTM Molar, 3M Deutschland GmbH) was temporarily filled in the access cavity for all groups. An intraoral periapical radiograph had been done immediately following root canal obturation by a Carestream RVG 5200 digital imaging system (Carestream Health Inc.). Every participant was instructed to return to the doctor for taking analgesics (ibuprofen 400 mg every 8 hours) to relieve the pain if needed and if severe pain persisted even after taking the prescribed analgesic or swelling appeared. At this point, similar to other patients in the trial, these patients were assessed again at 24, 48, and 72 hours and continued till the seventh day.

post operative evaluation The possibility of pain developing was explained to patients. After the root canal procedure was finished, postoperative pain was recorded through the VRS at 6h., 12h., 24h., 48h., and 72 hours and following one week. The VRS was a pain scale with pain scores (16) of none at all; the patient reported no discomfort (Vas score 0). Mild (Vas score 1), noticeable but not uncomfortable. Moderate (Vas score 2): uncomfortable but manageable. Severe (Vas score 3): significant discomfort that was difficult to tolerate. Every participant received a chart to document their level of discomfort following the procedure as well as how often they take analgesics postoperatively.

Statistical analysis: - The collected data will be, tabulated, and statistically analyzed using SPSS program (Statistical Package for Social Sciences) software version 23.0. Descriptive statistics will be done for numerical parametric data as mean±SD (standard deviation) and minimum & maximum of the range and for numerical non parametric data as median and 1st& 3rd inter-quartile range, while they will be done for categorical data as number and percentage. Inferential analyses will be done for quantitative variables using independent t-test in cases of two independent groups with parametric data and Mann Whitney U in cases of two independent groups with non-parametric data.

Inferential analyses will be done for qualitative data using Chi square test for independent groups. The level of significance will be taken at P value <0.050 is significant, otherwise is non-significant. The p-value is a statistical measure for the probability that the results observed in a study could have occurred by chance.

ELIGIBILITY:
Inclusion Criteria:

* solitary-rooted lower premolar teeth with acute irreversible pulpitis and apical periodontitis who were in the age range between 18 and 40 years old.
* Each patient received root canal treatment in one session.
* restorable teeth with a normal periodontal score index of less than two
* severe preoperative pain (Vas score 3)
* discomfort response on biting/mastication or percussion but no mobility.
* Discomfort response on palpation of surrounding tissue but with no intraoral swelling.
* Patients who stopped medications for the last 12 hours before the procedure
* The radiograph showed only normal or slight widening in the periodontal ligament space of the affected root.

Exclusion Criteria:

* patients with any serious systemic disease
* Patients under the age of eighteen or incapable of giving informed consent
* Patients over forty
* Patients with a mandibular premolar involving multiple canals or huge periapical pathosis
* Patients with severe preoperative pain on biting/mastication or percussion
* Mandibular premolar with open apices
* Mandibular premolar with periodontal involvement
* Retreated cases, sinus tract presence, and swelling of surrounding soft tissues
* patients who had been pregnant and allergic patients with local anesthetic agents

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
The Impact Of Different Final Irrigation Activation Techniques On Postoperative Pain | 6, 12, 24, 48, 72 hours and I week after completion of root canal treatment.
  Patients will be informed about the possible development of pain. Postoperative pain will be assessed using a VRS 6, 12, 24, 48, 72 hours and I week after completion of root canal treatment. The VRS consisted of a four-step pain scale using a continuous 0-3 point scale; No pain (0): the treated tooth felt normal. Patients did not have any pain or discomfort, mild (1): recognizable, not discomforting), moderate (2): discomforting, but bearable, and severe (3): considerable discomfort, difficult to bear.
  Each participant will be given a chart to record the level of postoperative pain and the frequency rate of the analgesic intake.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin T sobh, PHD, Principal Investigator — faculty of Dentistry , sinai university
Locations (1):
- Sinai University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No